CLINICAL TRIAL: NCT05874947
Title: Accuracy of Different Technologies for Dental Cast Digitization; CBCT Versus Desktop Optical 3D Scanner: An Observational Study
Brief Title: Accuracy of Different Technologies for Dental Cast Digitization; CBCT Versus Desktop Optical 3D Scanner
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Hamdy Mohammed Elfaramawy, Principal investigator, Cairo University
Other Study IDs: radiology1
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Evaluate and Compare the Accuracy of Digital Dental Models Generated From Plaster Casts by Two Different Scanning Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dental Cast Digitization techniques:(CBCT 3D model scanning module ): Scanning the plaster model using CBCT 3d model scanning module to generate a digital model
  Interventions: Device: linear measurement
- Dental Cast Digitization techniques :Desktop Optical 3D Scanner: Scanning the plaster model using Desktop Optical 3D Scanner to generate a digital model
  Interventions: Device: linear measurement
- plaster cast: linear measurments on the plaster cast as the gold standard (using the digital caliper )
  Interventions: Device: linear measurement

INTERVENTIONS:
Device: linear measurement — Linear measurements from digital caliper ,CBCT and EOS generated digital dental models

SUMMARY:
The objective of this study is to evaluate and compare the accuracy of digital dental models generated from plaster casts by two different scanning techniques including Cone Beam Computed Tomography (CBCT) and extraoral Scanner (EOS) .

The comparison between the two techniques is assessed by orthodontic arch space analysis using linear measurements for arch length and width .

ELIGIBILITY:
Inclusion Criteria:

* Patients with maxillary or mandibular complete permanent dentition
* Partially edentulous patients provided the dentition are complete from the first molar to the first molar.

Exclusion Criteria:

* Patients with fractured teeth, attrition and/or erosion affecting the anatomical points
* Patients having non-anatomic restorations that may alter cusp anatomy affecting the accuracy of measurements consequently.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Population selected for this study is any healthy male/female participant with complete set of non fractured maxillary or mandibular permanent teeth first molars included.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
Deviation of CBCT and extraoral scanner's measurements from gold standard in arch space analysis. | one year
  Evaluate and compare the accuracy of digital dental models generated from plaster casts by two different scanning techniques including Cone Beam Computed Tomography (CBCT) and extraoral Scanner (EOS).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry ,Cairo University, Cairo, Almanial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided